CLINICAL TRIAL: NCT00923650
Title: Informed Consent in Pediatric Phase I Cancer Trials
Brief Title: Informed Consent in Pediatric Cancer Trials
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090052; 09-C-0052; NCT00891410 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-02

CONDITIONS: Osteosarcoma; Ewing's Sarcoma; Neuroblastoma; Brain Tumors; Leukemia
Keywords: Informed Consent; Pediatric Phase I Clinical Trials; Assent; Questionnaires; Osteosarcoma; Ewing's Sarcoma; Neuroblastoma; Brain Tumors; Leukemia
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Neuroblastoma; Brain Neoplasms; Leukemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Informed consent is the process by which prospective participants in clinical trials learn about clinical research in order to decide whether they want to enroll in the study. It consists of meetings and discussions with the health care team.
* Phase I clinical trials are designed to determine what dose of an investigational agent is safe to administer to patients.

Objectives:

* To study communication, comprehension and decision-making during the informed consent process.
* To examine ethical, psychological, social, and educational issues regarding informed consent.
* To help researchers understand how to improve informed consent and education about clinical research.

Eligibility:

* Parents or guardians of children with cancer who are being considered for participation in phase I clinical trials
* Prospective patients for pediatric phase I clinical trials who are between 14 and 21 years of age.
* Members of the research team who obtain consent from patients and families for pediatric phase I clinical trials

Design:

* Research assistants observe and record the informed consent conference held with the research team and the parents and children.
* After the conference, the research assistant interviews the parents in a private area about their experience during the conference and their decision-making process. They are asked about their thoughts and opinions during the informed consent conference, including the decision-making process, communication and trust in the medical team.
* With their parent's permission, patients are interviewed privately to discuss their experience during the informed consent conference.
* After parents and patients have made their decision about participation in the study, they are interviewed again about how they made the decision, aspects of the communication during the conference, and how they feel about the doctor. This interview is also recorded.
* Parents may be contacted 6 months to 2 years from the time of their participation to be part of a parent advisory group about the informed consent process.

DETAILED DESCRIPTION:
Background:

* The clinical course and poor prognosis of children and adolescents eligible for pediatric phase I trials may increase the vulnerability of patients and their families and confound informed consent
* Physicians report a tension between presenting reasonable options and a truthful prognosis while maintaining hope.
* Research on the communication and decisions regarding participation in pediatric phase I trial is needed.

Objectives:

* The primary objective of this study is to understand communication, comprehension, and decision-making in Phase I childhood cancer trials (Specific Aim 1) by examining:

  * The way that phase I pediatric trials are presented (Aim 1 Hypothesis 1)
  * Whether and how alternatives (such as hospice) are introduced (Aim 1 Hypothesis 2)
  * What parents and children older than 14 years understand after the consent discussion (Aim 1 Hypothesis 3)
  * How the communication process influences parental comprehension and decision-making regarding participation of their child in a phase I study (Aim 1 Hypothesis 4)
  * How clinician-investigator perspectives may vary from that of the parent of a child participating in a phase I study (Aim 1 Hypothesis 5)
* Compare Phase I vs. Phase III pediatric cancer informed consent (Specific Aim 2) regarding:

  * Parental understanding of the scientific goals of the trial (Aim 2 Hypothesis 1)
  * Trust, decision making preferences, strength of recommendation by investigators interactivity as measured by number of parental questions, reasons for decisions, child's involvement, reading consent document, parental understanding of choice and trial design/purpose, disclosure of prognosis (Aim 2 Hypothesis 1-9)
  * Develop suggestions for interventions to improve informed consent in Phase I pediatric cancer trials through Parent Advisory Group on Informed Consent (PAGIC).(Specific Aim 3)

Eligibility:

* Parents or guardians of children and adolescents considering enrollment on Phase I Trials of anti-cancer agents, gene transfer or vaccine studies are eligible if the child or adolescent is less than 22yrs with diagnosed with a recurrent or refractory malignant solid tumor or leukemia.
* Participants must speak English or Spanish.
* Parents or guardians of children or adolescents who are newly diagnosed with cancer or previously participated in informed consent research are excluded.
* In addition, we plan to interview a smaller number of patients who are 14-21 years of age and who have participated in an informed consent conference for a Phase I cancer trial.

Design:

* Parents (n=132) of children or adolescents (age less than or equal to 21 years) who are being offered participation in a Phase I clinical trial for cancer will be sequentially recruited.
* The methods will include direct observation, digital recording of ICC, and questionnaires of parent/guardian, patients, and health care team members. Research Assistants (RAs) will be trained to observe and record all interactions between families and clinicians that relate to the Phase I clinical trial. Children over 14 years old will be interviewed using a separate instrument
* Data will be analyzed by quantitative and qualitative analytic methods. To assure 120 cases for analysis, the total accrual is 132 cases at six institutions, up to 100 will be accrued at the NCI.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Parent/Guardian:

  * Patient must be less than or equal to 21 years of age at the time of consent.
  * Parent/guardian must be considering having their child participate in a Phase I treatment trial
  * Parents must be able to speak English or Spanish
  * Must sign informed consent for participation in this study
* Patients greater than or equal to14 years of age and less than or equal to 18 years of age:

  * Must be considering participating in a Phase I treatment trial
  * Must be able to speak English or Spanish
  * Must assent for participation in this study
* Patients greater than or equal to 18 years old:

  * Must be considering participating in a Phase I treatment trial
  * Must be able to speak English or Spanish
  * Must sign informed consent for participation in this study, which will include consent to interview parent/guardian, if available
* Heath Care Team Members:

  * Must be greater than or equal to 18 years of age
  * Must speak English or Spanish
  * Must sign an informed consent document for participation in this study (written consent will be obtained annually for heath care team members)
  * Verbal assent to participate in each individual consent conference

EXCLUSION CRITERIA:

* Patients who are newly diagnosed who are being offered participation in a Phase I trial because no standard therapy exists for their disease
* Patients/Parents who have previously participated in informed consent research conducted by Cleveland Clinic Foundation Department of Bioethics
* Families who do not speak English or Spanish

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2008-12-09; Study Completion 2010-02-02

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Cleveland Clinic Foundation Childrens Hospital, Cleveland, Ohio

REFERENCES:
- [Background] Sunkel C, Cillero F, Armijo M. [2-(p-Acetamidophenyloxy)ethyl-o-acetoxybenzoate (eterilate). A new anti-inflammatory derived from acetylsalicylic acid. Synthesis and its physico-chemical properties]. Arch Farmacol Toxicol. 1978 Apr;4(1):153-5. No abstract available. Spanish. PMID 697385
- [Background] Lind SE. Can patients be asked to pay for experimental treatment? Clin Res. 1984 Oct;32(4):393-8. No abstract available. PMID 6509865
- [Background] Ting AT, Karnitz LM, Schoon RA, Abraham RT, Leibson PJ. Fc gamma receptor activation induces the tyrosine phosphorylation of both phospholipase C (PLC)-gamma 1 and PLC-gamma 2 in natural killer cells. J Exp Med. 1992 Dec 1;176(6):1751-5. doi: 10.1084/jem.176.6.1751. PMID 1281218